CLINICAL TRIAL: NCT03839901
Title: A Pilot Study to Investigate Two Different Physiotherapy Rehabilitation Programmes, to Treat the Conservatively Managed Scapholunate Instability.
Brief Title: Rehabilitation Programmes for Scapholunate Instability
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There were insufficient numbers recruited before the end of the student project
Sponsor: University of Bradford (Other)
Collaborators: Bradford Teaching Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS 218328
Record Dates: First submitted 2019-01-28; First posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Wrist Strain; Wrist Sprain; Scaphoid-Lunate Instability
Keywords: Scaphoid-Lunate; instability; wrist

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isometric training programme (Experimental): 'Home exercise programme' consisting of isometric exercises with participants followed up at week 1, 4, 6 and 8.
  Interventions: Other: Home exercise program
- isotonic training programme (Experimental): 'Home exercise programme' consisting of isotonic exercises with participants followed up at week 1, 4, 6 and 8.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Home exercise program — Home exercise programme with participants followed up at week 1, 4, 6 and 8.

SUMMARY:
Two different exercises approaches were tested in patients with Scapho-Lunate (SL) instability; one to strengthen the tendons in static positions and the other to strengthen the tendons whilst the wrist is moving.

DETAILED DESCRIPTION:
Scapho-Lunate (SL) instability is the most common form of wrist instability, but is complex to diagnose and is often missed entirely. The natural progression of SL instability has been suggested to lead to osteoarthritis. The management of SL instability can be broadly divided into conservative and surgical, with the former being the first option taken by most medical professionals, which primarily involves physiotherapy. The evidence base for physiotherapy management of SL instability is limited; however cadaver research has identified loading some of the wrist tendons may stabilise the scaphoid and lunate.There is currently no research as to whether this clinically makes any difference to the patients symptoms, or how to do it. This research therefore aimed to test the protocol and methods, and act as a platform for larger studies, to investigate this.

Two different exercises approaches were tested; one to strengthen the tendons in static positions and the other to strengthen the tendons whilst the wrist is moving.

ELIGIBILITY:
Inclusion Criteria:

* Ages eighteen to sixty,
* wrist pain,
* confirmed scapholunate ligament disruption on MRA or XR (partial or full),
* referred from orthopaedic wrist specialist,
* for conservative management,
* consent to trial.

Exclusion Criteria:

* Under eighteen or over sixty years,
* previous fracture,
* degenerative changes in the wrist,
* previous surgery,
* complex regional pain syndrome or diagnosis of rheumatological conditions,
* no wrist injection in preceding twelve months or other wrist conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Grip strength using E-link dynamometer | assessed at 0, 4 and 8 weeks
  change of grip strength from baseline change of 20% in kg considered signifcant

SECONDARY OUTCOMES:
numerical rating scale | assessed at 0, 4 and 8 weeks
  Pain scored on a numerical rating scale 0 (no pain) -10 (unbearable pain) Minimally Clinical Important Difference of 20mm
Patient Rated Wrist Evaluation | assessed at 0, 4 and 8 weeks
  Used Patient Rated Wrist Evaluation PRWE questionnaire (A score of 100 represents the worst functional score, whereas 0 represents no disability) with Minimally Clinical Important Difference of 14 points

CONTACTS AND LOCATIONS:
Locations (1):
- Bradford Royal Infirmary, Bradford, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No